CLINICAL TRIAL: NCT04306549
Title: Twenty-Four-Month Clinical Comparison of Two Bulk-Fill and Microhybrid Composite Restorations
Acronym: Clinical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: University of Beykent (Other); Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Emine Sirin Karaarslan, Assoc.Proffesor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/36
Record Dates: First submitted 2020-03-03; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Dental Restoration Failure of Marginal Integrity
Keywords: Clinical study; USPHS criteria; bulk-fill; resin composite; Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bulk-fill resin composite-sonic activated (Experimental): 5 mm bulk-filling without capping lightcured 40s
  Interventions: Other: Bulk-Fill and Microhybrid Composite Resins
- Bulk-fill resin composite (Experimental): 4 mm bulk-filling without capping lightcured 10s
  Interventions: Other: Bulk-Fill and Microhybrid Composite Resins
- Microhybrid resin composite (Experimental): 2 mm layers, lightcured 20s
  Interventions: Other: Bulk-Fill and Microhybrid Composite Resins

INTERVENTIONS:
Other: Bulk-Fill and Microhybrid Composite Resins — Clinical Comparison of Composite Restorations (Two Bulk-Fill and one Microhybrid Composite Resin) to the USPHS Criterias
  Other Names: Twenty-Four-Month Clinical Comparison of Two Bulk-Fill and Microhybrid Composite Restorations

SUMMARY:
ABSTRACT Objective The aim of this study was to evaluate the clinical performance of one microhybrid and two bulk-fill resin composites in Class II cavities for up to two years.

Materials and methods In total, 75 Class II restorations were made in 25 patients, using three restorative materials: two nanohybrid bulk-fill resin composites, Sonic Fill (SF) and x-tra fil (XF), and a microhybrid composite, Filtek Z-250 (FZ). The restorations were blindly evaluated by two examiners at baseline and at 6, 12, and 24 months, using U.S. Public Health Service (USPHS) criteria. The restoration groups for each category were compared using the Pearson chi-square test, and the Cochran Q-test was used to compare the changes across different time points within each restorative material (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* Patient in need of restoration of caries lesion (diagnosed with bitewing radiograph and clinical examination);
* teeth in need of restoration to be first or second molars or permanent premolars;
* at least three Class II restorations required in each patient and the number of restorations of each material to be equal in each patient;
* the antagonist and adjacent tooth in contact;
* pulp vitalized and free of painful symptoms; teeth involved not to have undergone direct pulp capping;
* no history of hypersensitivity in the teeth to be restored;
* permanent dentition;
* good oral health and absence of periodontal disease;
* patients not to have suffered from systemic diseases or allergies;
* absence of deleterious habits, xerostomia, and bruxism.

Exclusion Criteria:

* Fewer than 20 teeth;
* history of existing tooth sensitivity;
* known allergy to resin-based materials or any of the other materials used in this study;
* pregnancy or breastfeeding;
* chronic use of anti-inflammatory drugs, analgesic, and/or psychotropic drugs;
* non-vital teeth;
* abutment teeth for fixed or removable prostheses.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Clinical Acceptability | Twenty-Four-Month
  One week after restoration placement (baseline), patients were recalled and restorations were examined clinically. Direct clinical evaluation of restorations was performed using the USPHS criteria by two independent investigators using mirrors, probes, and bitewing radiographs and scored as Alpha, Bravo, or Charlie. Alpha corresponded to excellent, Bravo to clinically acceptable, and Charlie to clinically unacceptable results. Patients were recalled at 6, 12, and 24 months for assessments of the restorations, using the same criteria as at baseline. At each recall, the same two calibrated evaluators, who were blinded to the restoratives used for cavities and patients, examined the restorations. To ensure a double-blind study, the evaluators were not informed about which filling material had been used on which teeth.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: one year

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT04306549/Prot_SAP_000.pdf